CLINICAL TRIAL: NCT06467227
Title: EFFECTIVE AEROBIC EXERCISE TRAINING IN HEALTH AND CHRONIC DISEASE. Part I: A Demonstration of Practical Implications of Muscle Recruitment on Exposure to the Aerobic Training Stimulus in Healthy Individuals
Brief Title: Exposure to the Aerobic Training Stimulus in Healthy Individuals
Acronym: O2MVPaA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Park Healthcare Centre (Other)
Responsible Party: Principal Investigator, Roger Goldstein, Director, Program in Respiratory Rehabilitation, West Park Healthcare Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: O2MVPaA-RG2024
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: A prospective longitudinal, self-controlled, single-case repeated measures, randomized and counterbalanced cross-over experimental trial design, comparing cardiopulmonary response and endurance with different modes of exercise
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: exercise modality — exercise using legs and arms

SUMMARY:
Fitness is an important determinant for health and influenced by using large muscles. Muscles respond to training. We want to know if adding arm exercise to leg exercise can provide a better training session for healthy individuals. If the strategy shows promise for healthy people then it might work for people with lung disease who have trouble training because of difficulty breathing. The purpose of this first study is to evaluate, in healthy people, a unique approach to training by determining if adding arm exercise to leg exercise can be endured longer than leg exercise alone.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals

Exclusion Criteria:

* orthopedic or neurological condition that might affect the performance of the treadmill, arm or leg cycling
* have a symptomatic cardiac disease or undergone a recent surgical procedure that might affect the performance on an exercise test
* presence of any chronic respiratory condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
cycling endurance time | 30 minutes
  tolerance (time) of an individualized constant power endurance test

CONTACTS AND LOCATIONS:
Overall Officials: Roger Goldstein, Principal Investigator — West Park Healthcare Centre
Locations (1):
- Westpark Health Care Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No